CLINICAL TRIAL: NCT03850327
Title: BIO|CONCEPT.BIOMONITOR III
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RD020
Record Dates: First submitted 2019-02-11; First posted 2019-02-21 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2018-12

CONDITIONS: Atrial Fibrillation; Syncope; Tachyarrhythmia
Keywords: Implantable Cardiac Monitor
MeSH Terms: conditions — Atrial Fibrillation; Syncope; Tachycardia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BIOMONITOR III (Experimental)
  Interventions: Device: BIOMONITOR III

INTERVENTIONS:
Device: BIOMONITOR III — Patients with ICM indication receive a third-generation implantable cardiac monitor

SUMMARY:
The objective of the study is to confirm the safety and efficacy of the BIOMONITOR III system. Furthermore, the insertion procedure, the use and handling of the incision and insertion tools and the sensing quality of the BIOMONITOR III will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patient is at high risk of developing a clinically important cardiac arrhythmia; or Patient is undergoing investigation for symptoms such as palpitations, pre-syncope or syncope, that are suggestive of an underlying cardiac arrhythmia; or Patient is undergoing investigation for the detection of atrial fibrillation following cryptogenic stroke; or Patient is planned for AF ablative procedure or has already undergone an AF ablative procedure.
* Patient is able to understand the nature of study and has provided written informed consent.
* Patient is willing and able to perform all follow up visits at the study site.
* Patient is willing and able to use the CardioMessenger and accepts the BIOTRONIK Home Monitoring concept.

Exclusion Criteria:

* Patients implanted with ICD or pacemaker.
* Patient is pregnant or breast feeding.
* Patient is less than 18 years old.
* Patient is participating in another interventional clinical investigation
* Patient´s life-expectancy is less than 6 months.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-03-08 (Actual); Primary Completion 2019-10-06 (Actual); Study Completion 2019-10-06 (Actual)

PRIMARY OUTCOMES:
Adverse Events | 1 month
  (procedure / device related)
R-wave amplitude | 1 month

SECONDARY OUTCOMES:
Insertion procedure of the BIOMONITOR III by using the incision and insertion tools | At the day of insertion of the BIOMONITOR III
  Assessment of insertion procedure by using a questionaire about handling and time record.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier van den Brink, Dr., Principal Investigator — The Alfred Hospital, Melbourne, Australia
Locations (7):
- Australia (7):
  - HeartCare Partners - Wesley Testing, Auchenflower, Queensland
  - Bundaberg Cardiology, Bundaberg, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - HeartCare Victoria - Doncaster, Balwyn, Victoria
  - Mount Hospital, Perth, Western Australia
  - The Canberra Hospital, Canberra
  - The Alfred Hospital, Melbourne